CLINICAL TRIAL: NCT03734796
Title: The Study of High-sEnsitivity cArDiac Troponin I vaLues and Changes In diagNosis of suspEcted Acute Coronary Syndrome Patients in China
Brief Title: Hs-cTnI Diagnosis of NSTE-ACS Patients in China
Acronym: HEADLINES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: HEADLINES
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Non-ST-elevation Myocardial Infarction (NSTEMI)
Keywords: High-sensitive cardiac troponin; Non-ST-elevation Myocardial Infarction (NSTEMI); Chinese; Acute chest pain
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- suspected NSTEMI: Patients aged 18-75 years old and highly suspected NSTEMI without Left bundle branch block (LBBB) will be included. Patients will be excluded if who is STEMI, underwent surgical operation within four weeks, medium and several kidney dysfunction (Ccr<30ml/min), anemia, acute myocarditis, chronic cardiac dysfunction (NYHA III-IV), serious cardiac arrhythmias, with history of intravenous drug, oncosis and recent thrombolysis treatment, or pregnant.

SUMMARY:
This study is to validate 1-hour and 3-hours diagnostic strategy using Architect high-sensitivity cardiac troponin I (hs-cTnI) in Chinese patients with suspected Non-ST-elevation Myocardial Infarction (NSTEMI). The accuracy of 1-hour and 3-hours algorithm of NSTEMI using hs-cTnI assays will be evaluated in China emergency patients. This trail is going to determine the optimal diagnostic cut-off value of NSTEMI in Chinese population according to 24-hour or longer clinical diagnosis of MI in routine way.

DETAILED DESCRIPTION:
Cardiac Troponin is recommended as a preferred cardiac biomarker in third universal definition of myocardial infraction. The validated high-sensitive cardiac troponin I is also considered competent 1-hour algorithm to rule out and/ rule in NSTEMI in 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. However, the diagnostic threshold of 1-hour and 3-hour need more solid evidence in Chinese population. This study is to validate 1-hour and 3-hours diagnostic strategy using Architect high-sensitivity cardiac troponin I (hs-cTnI) in Chinese patients with suspected non-ST-elevation Myocardial Infarction (NSTEMI). The accuracy of 1-hour and 3-hours algorithm of NSTEMI using Architect hs-cTnI assays will be assessment in China emergency patients. This trail is going to determine the optimal diagnostic cut-off value of NSTEMI in Chinese population according to 24-hour or even longer clinical diagnosis of MI in routine way.

In primary phase of the present study, 400 patients with acute chest pain, who suspected NSTE-ACS, will be enrolled when visiting emergency department of Fuwai hospital. In subsequent study, multi center emergency department in China plan to recruit 2000 patients suspected NSTE-ACS. The inclusion and exclusion criteria had been described in the following eligibility part. All recruited patients undergo an initial clinical assessment including clinical history, physical examination, 12-lead ECG monitoring, routine blood measurements and echocardiogram. The blood samples of patients will be collected according to standard biobank protocol. Cardiac troponin I, CK-MB and myoglobin will be measured at presentation, 1-hour, 3-hours and 12-hours employing contemporary cTnI and high-sensitive cTnI, respectively.

The diagnosis of each enrolled patient will be made according to routine clinical approach and 1-hour and 3-hours clinical approach, respectively. The routine clinical diagnosis will be made by cardiologist panel according to third universal definition of myocardial infraction through reviewing all available medical records. The NSTEMI diagnosis depended on Architect hs-cTnI assessment will be made a senior cardiologist according to 1-hour and 3-hours clinical approach recommended by 2015 ESC guidelines for the management of NSTEMI. When there was disagreement about the diagnosis, cases were reviewed and adjudicated in conjunction with a third senior cardiologist.

Finally, statistical expert will evaluate the diagnostic performance of 1-hour and 3-hours clinical approach and diagnostic threshold of NSTEMI when the new hs-cTnI employed.

ELIGIBILITY:
Inclusion Criteria:

* 18-75y;
* highly suspected NSTEMI;
* ECG results without ST-segment elevation;
* without new Left bundle branch block (LBBB) ;

Exclusion Criteria:

* STEMI;
* underwent major surgical operation or injury within four weeks;
* medium and several kidney dysfunction (Ccr<30ml/min);
* anemia(Hb<90g/L);
* acute myocarditis;
* chronic cardiac dysfunction (NYHA III-IV);
* serious cardiac arrhythmias;
* Have had similar symptoms and treatment with thrombolysis before one month;
* history of intravenous drug;
* history of oncosis;
* pregnant;
* even recruited;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In primary phase of the present study, 400 patients with acute chest pain, who suspected NSTEMI, will be enrolled when visiting emergency department of Fuwai hospital. In subsequent study, multi center emergency department in China plan to recruit 2000 patients suspected NSTEMI. Patients aged 18-75 years old and highly suspected NSTEMI without Left bundle branch block (LBBB) will be included. Patients will be excluded if who is STEMI, underwent surgical operation within four weeks, medium and several kidney dysfunction (Ccr<30ml/min), anemia, acute myocarditis, chronic cardiac dysfunction (NYHA III-IV), serious cardiac arrhythmias, with history of intravenous drug, oncosis and recent thrombolysis treatment, or pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Myocardial Infarction | 0 - 72 hour
  Number of Participants with NSTEMI

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liang, MD, Study Chair — Department of Emergency Medicine, State Key Laboratory of Cardiovascular Disease National Center for Cardiovascular Diseases & Fuwai Hospital Peking Union Medical College & Chinese Academy of Medical Sciences; Zhou Zhou, MD, PhD, Study Chair — Center of Laboratory Medicine Beijing Key Laboratory for Molecular Diagnostics of Cardiovascular Disease State Key Laboratory of Cardiovascular Disease National Center for Cardiovascular Diseases & Fuwai Hospital Peking Union Medical College & Chinese Aca
Locations (1):
- Yan Liang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No